CLINICAL TRIAL: NCT05444803
Title: Comparison of Femoral Nerve Block Versus Peri-capsular Nerve Group Block for Analgesia During Positioning for Spinal Anesthesia in Patients With Hip Fracture
Brief Title: Femoral Nerve Block vs Peri-capsular Nerve Group Block for Hip Fracture Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: safa1
Record Dates: First submitted 2022-06-20; First posted 2022-07-06 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-06

CONDITIONS: Spinal Anesthesia; Analgesia; Hip Fractures
MeSH Terms: conditions — Agnosia; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral nerve block group (Other): Thirty minutes before the placement of spinal block, patients will be receive a femoral nerve block with Bupivacaine.
  Interventions: Other: femoral nerve block
- Peri-capsular nerve group block group (Other): Thirty minutes before the placement of spinal block, patients will be receive a peri-capsular nerve group block with Bupivacaine.
  Interventions: Other: peri-capsular nerve group block

INTERVENTIONS:
Other: femoral nerve block — Patients will be performed a femoral nerve block using bupivacaine thirty minutes before the performing of spinal block.
  Arms: Femoral nerve block group
Other: peri-capsular nerve group block — Patients will be performed a peri-capsular nerve group block using bupivacaine thirty minutes before the performing of spinal block.
  Arms: Peri-capsular nerve group block group

SUMMARY:
The purpose of the study is to compare the analgesic efficacy of femoral nerve block and peri-capsular nerve group block administered before spinal anesthesia for positioning to spinal anaesthesia in patients undergoing surgery for hip fracture and to evaluate the efficacy for postoperative analgesia

DETAILED DESCRIPTION:
Spinal anesthesia is commonly used in patients undergoing hip fracture surgery. However the procedure of patient positioning to perform a spinal block is painful and may require the administration of IV analgesics or some regional anesthesia techniques such as femoral nerve block, fascia-iliaca compartment block, peri-capsular nerve group block. At the study, the investigators aimed to compare analgesic efficacy of femoral nerve block and peri-capsular nerve group block administered before spinal anesthesia for positioning to spinal anaesthesia in patients undergoing surgery for hip fracture and to evaluate the efficacy for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients with hip fracture scheduled for surgery under spinal anesthesia.

Exclusion Criteria:

* hemorrhagic diathesis,
* peripheral neuropathy,
* allergy to local anesthetics,
* mental disorders,
* use of analgesics for 8 h before the performance of spinal block

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Rate of pain scores assessed by Numerical rating Score Scale during positioning for spinal anesthesia | 30 minutes
  Pain scores will be assessed by Numerical Rating Scale (NRS) scores (from 0=no pain to 10=maximum possible pain).

SECONDARY OUTCOMES:
Rate of pain scores at rest | 30 min
  Pain scores will be assessed by Numerical Rating Scale (NRS) scores from 0 (no pain) to 10 (maximum possible pain) at rest before and 30 min after the block performance.
Rate of pain scores on passive limb lifting | 30 min
  Pain scores will be assessed by Numerical Rating Scale (NRS) scores from 0 (no pain) to 10 (maximum possible pain) on passive limb lifting before and 30 min after the block performance.
rate of postoperative pain scores | 24 hours
  Pain scores will be assessed by Numerical Rating Scale (NRS) scores from 0 (no pain) to 10 (maximum possible pain).at 6, 12, 24 hours postoperatively.
Amount of postoperative analgesic consumption | 24 hours
  Postoperative analgesic consumption will be recorded for postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Safa Eroglu, M.D., Principal Investigator — Antalya Traning and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)